CLINICAL TRIAL: NCT02581488
Title: Clinical Outcomes for Diabetic Foot Ulcers Treated With Clostridial Collagenase (SANTYL®) Ointment or With a Comparator Product Containing Silver
Brief Title: Use of Santyl in Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017-101-09-035
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Foot; Foot Ulcer, Diabetic
Keywords: Diabetes; diabetic foot ulcer; foot sore; type 2 diabetes; type 1 diabetes; neuropathy; DFU
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Santyl (Experimental): Collagenase ointment applied topically once per day for up to six weeks.
  Interventions: Biological: Santyl
- Product containing silver (Active Comparator): Products containing silver will be applied per Investigator instructions and instructions for use/package insert for up to six weeks.
  Interventions: Other: Product containing silver

INTERVENTIONS:
Biological: Santyl
  Arms: Santyl
Other: Product containing silver — Silver product not specified by the protocol; Investigators choose the appropriate silver containing product for each diabetic foot ulcer
  Arms: Product containing silver

SUMMARY:
This study is designed to test the hypothesis that daily treatment of diabetic foot ulcers with an enzymatic debriding agent, SANTYL, for up to 6 weeks will result in more rapid decrease in ulcer area than diabetic foot ulcers treated with a topical treatment containing silver. After meeting study criteria, participants will be randomly assigned to apply SANTYL or a topical treatment containing silver to their to foot ulcer for up to 6 weeks. At the end of 6 weeks, participants will be followed for an additional 4 weeks to examine the outcome of the study treatment.

DETAILED DESCRIPTION:
The objectives of this study were to compare outcomes of diabetic foot ulcers (DFUs) treated with SANTYL or silver-containing products, both in combination with sharp debridement as needed. One hundred two subjects with qualifying DFUs were randomized to daily treatment with either SANTYL or a silver-containing product for 6 weeks followed by a 4 -week follow-up period. The primary outcome was the mean percent reduction in DFU area. A secondary outcome was the incidence of ulcer infections between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
2. Eighteen (18) years of age or older, of either sex, and of any race or skin type.
3. Willing and able to make all required study visits.
4. Able to follow instructions and perform the dressing changes at home or have a caregiver who can perform the dressing changes according to the protocol.
5. Willing to use an appropriate off-loading device to keep weight off of foot ulcers.
6. An ulcer present on any part of the plantar surface of the neuropathic foot or hallux which is 0.5 cm2 - 10 cm2 inclusive (as measured at the Screening Visit using the ARANZ Silhouette imaging device). The target ulcer duration must be ≥ 6 weeks but not more than 52 weeks (12 months) as documented in the subject's history or by subject report of onset, and which requires debridement.
7. Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.70 and ≤ 1.20. If ABI > 1.2, perfusion at or near the site of the ulcer should be confirmed; the foot is warm to the touch and has palpable pulses.
8. Separation of at least 5 cm (closest ulcer edge to other closest ulcer edge) if ≥ 2 ulcers are present as measured using the ARANZ Silhouette imaging device.
9. Diabetes mellitus (Type 1 or 2) requiring insulin or oral/injectable medications to control blood glucose levels.
10. Target ulcer is not infected based on clinical assessment.

Exclusion Criteria:

1. Contraindications or hypersensitivity to the use of clostridial collagenase or products containing silver.
2. Participation in another clinical trial within thirty (30) days of Visit 1, or planned participation overlapping with this study.
3. Bleeding disorder that would preclude sharp debridement during the study.
4. Active cellulitis of the target ulcer, lymphangitic streaking, deep tissue abscess, gangrene, or infection of muscle, tendon, joint or bone.
5. Infection with systemic toxicity or metabolic instability (e.g., fever, chills, tachycardia, hypotension, confusion, vomiting, leukocytosis, acidosis, severe hyperglycemia, azotemia).
6. A target ulcer which involves the underlying tissues of tendon, muscle, or bone.
7. Diagnosis of chronic granulomatous disease, leukocyte adhesion defects, or severe neutropenia.
8. Current treatment (at the time of the Screening Visit) with any of the following:

   * Systemic corticosteroids. If corticosteroid treatment was for ≥ 10 days, there must be a 1 week interval between discontinuation and screening.
   * Immunosuppressive agents
   * Chemotherapeutic agents
   * Antiviral agents
   * Systemic antibiotic therapy (for any reason) or topical antibiotic treatment of the target ulcer
9. Treatment of target ulcer with bioactive therapies within 1 month of screening:

   * Platelet-derived growth factor (e.g., Regranex®)
   * Living skin equivalent (e.g., Apligraf®)
   * Dermal substitute (e.g., Dermagraft®, Integra®, Oasis®, etc.)
   * Amniotic membrane products (e.g., EpiFix®, Grafix®, etc.)
10. Prior treatment of target ulcer for any length of time with clostridial collagenase ointment (SANTYL®).
11. Radiation therapy to the target lower extremity within 30 days prior to screening.
12. Medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.
13. Blood counts and blood chemistry values as follows:

    * Alanine aminotransferase (ALT) > 3x upper limit of normal
    * Aspartate aminotransferase (AST) > 3x upper limit of normal
    * Gamma Glutamyl Transferase (GGT) > 2.5x upper limit of normal
    * Serum albumin < 2.0 g/dL • Pre-albumin levels of < 10 mg/dL
    * Alkaline phosphatase > 500 U/L • Serum total bilirubin > 3.0 mg/dL
    * Serum BUN > 75 mg/dL • Serum creatinine > 4.5 mg/dL
    * HbA1c > 12% • Hemoglobin (Hgb) < 8.0 g/dL
    * WBC < 2.0 x 109/L • Absolute neutrophil count < 1.0 x 109/L
    * Platelet count < 50 x 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Eichelkraut, Study Chair — Smith & Nephew, Inc.
Locations (13):
- United States (11):
  - Sylmar, California
  - Melbourne, Florida
  - Baltimore, Maryland
  - Las Vegas, Nevada
  - York, Pennsylvania
  - Fort Worth, Texas
  - McAllen, Texas
  - St. George, Utah
  - Harrisonburg, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
- Canada (2):
  - Hamilton, Ontario
  - Boucherville, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Santyl: Collagenase ointment applied topically once per day for up to 6 weeks.
- Product Containing Silver: Products containing silver was applied per Investigator instructions and instructions for use/package insert for up to 6 weeks. Silver product was not specified by the protocol; Investigators chose the appropriate silver containing product for each diabetic foot ulcer.
Period: Overall Study
Arm/Group | Santyl | Product Containing Silver
Started | 51 | 51
Completed | 42 | 40
Not Completed | 9 | 11
Not completed — Adverse Event | 6 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-Compliance | 1 | 0
Not completed — Protocol Violation | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Santyl | Product Containing Silver | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (13.1) | 57.6 (10.8) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 42 | 36 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 37 | 35 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 47 | 47 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 10 | 10 | 20
  United States | 41 | 41 | 82
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (7.7) | 33.6 (6.3) | 34 (7.0)
Height [Mean (Standard Deviation); unit: inches] | 69.6 (3.2) | 68.8 (3.8) | 69.2 (3.5)
Weight [Mean (Standard Deviation); unit: lbs] | 237.6 (56.7) | 226.6 (49.1) | 232.1 (53.0)
Ankle Brachial Index [Mean (Standard Deviation); unit: ABI ratio (mmHg/mmHg)] — The Ankle-Brachial Index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachial). Lower values represent a worse outcome, indicating peripheral artery disease (PAD).
  ABI = Ankle Systolic Pressure (mmHg) / Arm Systolic Pressure (mmHg)
  Range of Scores based on American Diabetes Association Guidelines:
  ABI Value, PAD Severity; >1.30, Poorly Compressible; 0.91 - 1.30, Normal; 0.70 - 0.90, Mild; 0.40 - 0.69, Moderate; <0.40, Severe
  ABI ratio (mmHg/mmHg) | 1 (0.1) | 1 (0.2) | 1 (1)
Target Ulcer Area [Mean (Standard Deviation); unit: cm^2] | 1.6 (1.8) | 1.7 (2.0) | 1.6 (1.9)
Foot Perfusion [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0
  No | 3 | 6 | 9
  N/A, ABI not > 1.2 | 48 | 45 | 93
Target Ulcer Location [Count of Participants; unit: Participants]
  Forefoot | 33 | 42 | 75
  Hallux | 12 | 4 | 16
  Heel | 3 | 4 | 7
  Medial Forefoot | 2 | 1 | 3
  Lateral Heel | 1 | 0 | 1
Ulcer Duration [Mean (Standard Deviation); unit: days] | 106.8 (75.2) | 118.1 (77.7) | 112.4 (76.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Ulcer Area From Baseline to the End of the Treatment.
Description: Ulcer area was measured using the ARANZ Silhouette digital imaging and measurement device.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of change from baseline (cm2)
Arm/Group | Santyl | Product Containing Silver
Number analyzed (Participants) | 51 | 51
percentage of change from baseline (cm2) | 57.6 (53.1) | 41.3 (58.3)

2. Secondary Outcome: Target Ulcer Infection Rates in Each Treatment Group During the Treatment Period as Determined by Investigator-reported Adverse Events
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Santyl | Product Containing Silver
Number analyzed (Participants) | 51 | 51
Participants | 5 | 11

3. Other Pre Specified Outcome: Time to Closure for Ulcers Achieving Closure in Treatment Period
Description: Days to closure for ulcers that closed by end of treatment period.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Santyl | Product Containing Silver
Number analyzed (Participants) | 51 | 51
days | 31.1 (9) | 37.1 (7.7)

4. Other Pre Specified Outcome: Time to Closure for Ulcers Achieving Closure by End of Follow-up
Description: Days to closure for ulcers that closed by end of follow-up period.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Santyl | Product Containing Silver
Number analyzed (Participants) | 51 | 51
days | 43.0 (18.6) | 50.8 (14.6)

5. Post Hoc Outcome: Incidence of Debridements During Treatment Period
Description: Number of debridements performed during the treatment period by treatment group.
Time Frame: 6 weeks
Measure: Number; unit: occurences
Arm/Group | Santyl | Product Containing Silver
Number analyzed (Participants) | 51 | 51
occurences | 305 | 272

ADVERSE EVENTS:
Time Frame: 14.5 months
Description: Adverse events were coded using Medical Dictionary for Regulatory Activities (MedDRA) adverse event dictionary. The frequency of treatment-emergent adverse events (TEAE) was calculated for each body system, by preferred term, by treatment group, for number of subjects, and the proportion reporting the event for the safety population (SAF).
Arm/Group | Santyl | Product Containing Silver
All-Cause Mortality (participants affected / at risk) | 1/51 | 1/51
Serious Adverse Events (participants affected / at risk) | 5/51 | 8/51
Other Adverse Events (participants affected / at risk) | 25/51 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=51) | Product Containing Silver (N=51)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pyelonephritis acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Santyl (N=51) | Product Containing Silver (N=51)
Blister (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 9 (9)
Diabetic foot (Infections and infestations) | 4 (6) | 7 (9)
Skin abrasion (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Wound infection (Infections and infestations) | 5 (5) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI to submit results for proposed publication/presentation to the sponsor no later than 90 days prior to the submission. Sponsor to reply within 60 days. Submission of publication/presentation may be delayed an additional 6 months to permit filing of appropriate patent applications. If a multicenter publication is not submitted within 24 months of the conclusion of the study, the Investigator may publish individual site results after review by sponsor.